CLINICAL TRIAL: NCT00261599
Title: A Phase 3, Randomized, Double-Blind, Dose-Controlled Study to Assess the Efficacy and Safety of AQUAVAN® (Fospropofol Disodium) Injection for Minimal to Moderate Sedation in Patients Undergoing Colonoscopy
Brief Title: An Effectiveness and Safety Study of AQUAVAN® Injection (Fospropofol Disodium) for Sedation During Colonoscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3000-0522; MGI 3000-0522
Record Dates: First submitted 2005-12-01; First posted 2005-12-05 (Estimated); Last update posted 2008-11-07 (Estimated); Status verified 2008-11

CONDITIONS: Conscious Sedation
Keywords: Colonoscopy; Sedation; AQUAVAN; Fospropofol disodium; Colon polyps; Endoscopic outcomes; Endoscopic sedation; Endoscopy
MeSH Terms: conditions — Colonic Polyps | interventions — fospropofol; Injections

INTERVENTIONS:
Drug: AQUAVAN® (fospropofol disodium) Injection
Drug: Midazolam HCI

SUMMARY:
Very often patients receive medication before a diagnostic procedure, like a colonoscopy, to help them relax and stay calm during the procedure. This is called procedural or minimal-to-moderate sedation. One product used for sedation is called propofol. AQUAVAN (fospropofol disodium) is made as a water soluble form of propofol allowing for rapid sedation during the entire procedure. This study is designed to test AQUAVAN for sedation during colonoscopy procedures.

DETAILED DESCRIPTION:
This is a phase 3, randomized, double-blind, dose-controlled study designed to evaluate the efficacy and safety of a moderate dose of AQUAVAN compared to a subtherapeutic dose of AQUAVAN,both following pretreatment with an analgesic fentanyl, in patients who are undergoing elective colonoscopy. A group of patients will receive midazolam as a reference therapy.

Following completion of pre-procedure assessments, patients will be randomly assigned to 1 of 3 treatment groups at a 2:3:1 (AQUAVAN initial dose 1 [subtherapeutic dose]:AQUAVAN initial dose 2 [moderate dose]: initial Midazolam Reference Dose) allocation ratio on the day of the scheduled procedure.

A person skilled in airway management and authorized by the facility in which the colonoscopy is performed (such as a respiratory therapist, a study nurse, or a clinician) must be immediately available during the conduct of the study. All patients will be placed on supplemental oxygen via nasal cannula (4 L/min), and an ECG monitor, pulse oximeter, and blood pressure monitor will be attached prior to administration of study medication. All patients will receive an injection of analgesic pretreatment followed by the administration of study medication. This protocol recognized 2 distinct phases of sedation: Sedation Initiation and Sedation Maintenance. Assessments will be made to evaluate the patients for levels of sedation, clinical benefit of sedation, and adverse events. Blood samples will be collected for PK analysis.

ELIGIBILITY:
* Number of patients/site: Approximately 300 patients at up to 30 sites will be randomized into this study.
* Study Country Location: United States

Inclusion Criteria:

1. Patient must be able to understand required assessments and procedures.
2. Patient provides signed/dated Informed Consent and Health Insurance Portability and Accountability Act of 1996 (HIPAA) authorization after receiving a full explanation of the extent and nature of the study.
3. Patient must be at least 18 years of age at the time of screening.
4. If female, patient must be surgically sterile, postmenopausal, or not pregnant or lactating and must have been using an acceptable method of birth control for at least 1 month prior to dosing, with a negative urine pregnancy test result at screening and pre-dose.
5. Patient meets American Society of Anesthesiologists (ASA) Physical Classification System status of P1 to P4.

Exclusion Criteria:

1. Patient has a history of allergic reaction or hypersensitivity to any anesthetic agent, opioid, or benzodiazepine.
2. Patient does not meet nils per os (NPO) status per ASA guidelines or institution's guideline.
3. Patient has a Mallampati Classification Score of 4; OR a Mallampati Classification Score of 3 AND a thyromental distance ≤4 cm, or for any other reason has a difficult airway, in the opinion of the Investigator.
4. Patient has an abnormal, clinically significant 3-lead ECG finding at predosing period Day 0.
5. Patient has participated in an investigational drug study within 1 month prior to study start.
6. Patient is unwilling to adhere to pre- and postprocedural instructions.
7. Patient for whom the use of fentanyl citrate injection (fentanyl) is contraindicated.
8. Patient for whom the use of midazolam HCl injection (midazolam) is contraindicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2006-03; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Sedation Success - 3 consecutive modified OAA/S scores of ≤4 after administration of sedative medication AND completing the procedure without requiring the use of alternative sedative medication AND without requiring manual or mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: James Jones, MD, PharmD, Study Director — Eisai Inc.
Locations (20):
- United States (20):
  - Clinical Research Associates, Huntsville, Alabama
  - UCSF-Fresno/University Medical Center, Fresno, California
  - Borland-Groover Clinic, Jacksonville, Florida
  - Rockford Gastroenterology Associates, Rockford, Illinois
  - Welborn Clinic, Evansville, Indiana
  - Indiana University Medical Center/Clarian Health Partner, Indianapolis, Indiana
  - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Maryland Digestive Diseases Center, Laurel, Maryland
  - Shah Associates, Prince Frederick, Maryland
  - Oakland Colon & Rectal Associates, Royal Oak, Michigan
  - Center for Digestive Health, Troy, Michigan
  - Gastrointestinal Associates, PA, Jackson, Mississippi
  - Research Associates of New York (New York Gastroenterology Associates), New York, New York
  - Asheville Gastroenterology Associates, Asheville, North Carolina
  - WestHills Gastroenterology Associates, Portland, Oregon
  - Memphis Gastroenterology Group, PC, Germantown, Tennessee
  - Gastrointestinal Institute, Nashville, Tennessee
  - Alamo Research Center, San Antonio, Texas
  - Spokane Digestive Disease Center, Spokane, Washington
  - Wisconsin Center for Advance Research, Milwaukee, Wisconsin